CLINICAL TRIAL: NCT06780189
Title: Investigation of the Effects of Passive Smoking on Vital Signs, Motor Activity Levels, and Agitation Severity in Children Undergoing Tooth Extraction With Sedation
Brief Title: The Effects of Passive Smoking on Vital Signs, Anxiety, and Recovery Times in Children Undergoing Primary Tooth Extraction Treatment Under Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Elif Buse Kaplan, Research Assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/387
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Dental Sedation; Passive Smoking
Keywords: primary tooth; passive smoking; Tooth extraction; dental sedation
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individuals with a daily cigarette consumption of fewer than 10 cigarettes. (Experimental)
  Interventions: Procedure: Tooth Extraction and Post-Procedure Monitoring Under Sedation in Children Exposed to Passive Smoking
- Individuals who consume between 10 and 20 cigarettes per day (Experimental)
  Interventions: Procedure: Tooth Extraction and Post-Procedure Monitoring Under Sedation in Children Exposed to Passive Smoking
- Individuals who consume more than 20 cigarettes per day. (Experimental)
  Interventions: Procedure: Tooth Extraction and Post-Procedure Monitoring Under Sedation in Children Exposed to Passive Smoking
- Individuals who do not smoke (Active Comparator)
  Interventions: Procedure: Tooth Extraction and Post-Procedure Monitoring Under Sedation in Children Not Exposed to Passive Smoking

INTERVENTIONS:
Procedure: Tooth Extraction and Post-Procedure Monitoring Under Sedation in Children Exposed to Passive Smoking — This study is designed to evaluate the relationship between passive smoking and the vital parameters of children undergoing deep sedation. Additionally, the study aims to comprehensively assess and document the entire treatment process from start to finish by using the RASS, MASS, and PAED scales for postoperative evaluation.
  Arms: Individuals who consume between 10 and 20 cigarettes per day; Individuals who consume more than 20 cigarettes per day.; Individuals with a daily cigarette consumption of fewer than 10 cigarettes.
Procedure: Tooth Extraction and Post-Procedure Monitoring Under Sedation in Children Not Exposed to Passive Smoking — This study is designed to measure the differences in vital parameters of children undergoing deep sedation who are not exposed to passive cigarette smoke at home. Furthermore, the study aims to comprehensively evaluate and document the entire treatment process from start to finish using the RASS, MASS, and PAED scales for postoperative assessment.
  Arms: Individuals who do not smoke

SUMMARY:
The aim of this clinical study is to evaluate the effects of passive smoking on the vital parameters of children undergoing primary tooth extraction under sedation and to assess their anxiety levels throughout the process until discharge.

The main questions it aims to answer are:

1. Do the vital parameters of children who are passive smokers differ from those of non-passive smokers under sedation?
2. Does the amount of smoking by family members influence the child's vital parameters?
3. Does passive smoking affect recovery and awakening times following sedation?
4. Does passive smoking impact the anxiety levels of children during the period leading up to discharge?

Participans:

* Children aged between 4 and 6 years,
* Children with an ASA score of 1,
* Children with a Frankl score of 4, 5, or 6,
* Children with an indication for primary tooth extraction,
* Parents/guardians who do not use electronic cigarettes.

DETAILED DESCRIPTION:
Sample Size Calculation and Study Design

The sample size for this study was calculated based on the article by A.C. Torun et al. (1), titled "Sedative - Analgesic Activity of Remifentanil and Effect of Preoperative Anxiety on Perceived Pain in Outpatient Mandibular Third Molar Surgery." According to this reference, the minimum required sample size was determined to be 64, with a 95% confidence interval and 5% sensitivity. A total of 100 children were included in the study, of whom 36 were classified as non-passive smokers and 64 as passive smokers.

Inclusion Criteria

Participants included in the study must meet the following criteria:

* Children aged between 4 and 6 years,
* Children with an ASA physical status classification of 1,
* Children scoring 1 or 2 on the Frankl Behavior Scale,
* Children with an indication for primary tooth extraction.

Evaluation Parameters

1. Assessment of Passive Smoking:

   Before the sedation procedure, parents/guardians will complete a questionnaire to determine the child's exposure to passive smoking.
2. Monitoring of Vital Parameters:

   During the sedation procedure, all patients will be connected to a monitoring device to record their vital parameters.
3. Assessment During and After Sedation:

   * Richmond Agitation-Sedation Scale (RASS): This scale will be applied during the sedation procedure and for 5 minutes after the procedure is completed.
   * Modified Aldrete Score (MASS): This scale will be used to measure recovery time.
   * Pediatric Anesthesia Emergence Delirium (PAED) Scale: Starting from the moment the patient regains consciousness, scores will be recorded every 5 minutes.

Outcome Measurement

The data obtained from the questionnaires, monitoring devices, and applied scales will be analyzed to evaluate the effects of passive smoking on sedation outcomes, recovery times, and emergence behaviors. All measurements will be conducted with consistency and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 and 6 years,
* Children classified as ASA 1,
* Children scoring 1 or 2 on the Frankl Behavior Scale,
* Children who are uncooperative for tooth extraction in the pediatric dentistry clinic,
* Children with an indication for primary tooth extraction,
* Parents/guardians of Turkish origin,
* Families who provide consent to participate in the study.

Exclusion Criteria:

* Children classified as ASA 2,3, 4, 5, or 6,
* Children scoring 3 or 4 on the Frankl Behavior Scale,
* Children younger than 4 years or older than 6 years,
* Children with acute apical abscess or cyst in the tooth scheduled for extraction,
* Children with an indication for permanent tooth extraction,
* Parents/guardians who use electronic cigarettes,
* Parents/guardians undergoing nicotine replacement therapy,
* Parents/guardians who are not of Turkish origin,
* Families who do not wish to participate in the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation level | Start Time: Before the administration of sedative drugs. End Time: At the completion of the tooth extraction procedure under deep sedation.
  Oxygen saturation is a parameter that represents the percentage of oxygen bound to hemoglobin molecules in arterial blood. It is a critical physiological indicator that reflects whether sufficient oxygen is being transported to the body's tissues. Normal oxygen saturation levels typically range between 95% and 100%, while levels below this range are referred to as hypoxemia, indicating a deficiency in oxygen supply. Oxygen saturation is commonly measured using a non-invasive method known as pulse oximetry.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayıs University, Samsun, Atakum
  - Ondokuz Mayıs Üniversity Facult of Dentistry, Samsun, Atakum

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code